CLINICAL TRIAL: NCT04505891
Title: Enhanced Kidney Follow-up for AKI Survivors in Care Transitions (The ACT Study): Impact on Patient Reported Outcomes
Brief Title: Enhanced Kidney Follow-up for AKI Survivors in Care Transitions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erin Barreto, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-004204
Record Dates: First submitted 2020-08-04; First posted 2020-08-10 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury
Keywords: transitions of care; education; patient reported outcomes; chronic kidney disease; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention)
- Education alone (Active Comparator)
  Interventions: Behavioral: Education
- Education and follow-up (Active Comparator)
  Interventions: Behavioral: Education and follow-up

INTERVENTIONS:
Behavioral: Education — Kidney health education will be delivered prior to discharge by trained nurse educators.
  Arms: Education alone
Behavioral: Education and follow-up — In patients allocated to the education and follow-up arm, education along with a a post-discharge healthcare visit from a multidisciplinary care team will be performed.
  Arms: Education and follow-up

SUMMARY:
The purpose of this study is to assess the ability of education and outpatient kidney care follow-up in order to improve patient knowledge about acute kidney injury (AKI).

ELIGIBILITY:
Inclusion Criteria:

* KDIGO Stage 3 AKI
* Primary care provider at Mayo Rochester.

Exclusion Criteria:

* Patient with need for dialysis at discharge from hospital or hospice.
* Enrolled in the Primary Care Transition Program.
* Non-English speaking.
* Cognitive impairment.
* Dementia.
* Mini-Cog score of less than 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Modified Kidney Knowledge Survey (mKIKS) | 14-days after last study contact
  Assesses participants' objective knowledge about AKI causes, risk factors, and management. The minimum score is 0, maximum score is 15, higher scores indicate greater knowledge.

SECONDARY OUTCOMES:
Brief health literacy screen | 30-days post hospitalization
  A 4-item tool to assess health literacy. Minimum score of 0, maximum score 20, higher scores indicate higher health literacy
Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health 10 | 30-days post hospitalization
  Based on the provided responses, an overall summary score, and two subset scores - Global health physical and Global health mental can be calculated. Raw summed score are converted into T-scores. Higher scores indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Erin F Barreto, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] May HP, Herges JR, Anderson BK, Hanson GJ, Kashani KB, Kattah AG, Cole KC, McCoy RG, Meade LA, Rule AD, Schreier DJ, Tinaglia AG, Barreto EF; ACT Study Group. Posthospital Multidisciplinary Care for AKI Survivors: A Feasibility Pilot. Kidney Med. 2023 Oct 5;5(12):100734. doi: 10.1016/j.xkme.2023.100734. eCollection 2023 Dec. PMID 37964784
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials